CLINICAL TRIAL: NCT04563871
Title: A Phase II, Open-label, Single-arm, Multicenter, Efficacy and Safety of 80mg Osimertinib in Patients With Leptomeningeal Metastases(LM) Associated With EGFR Mutation-positive Non-small Cell Lung Cancer(NSCLC)
Brief Title: Efficacy and Safety of 80mg Osimertinib in Patients With Non-small Cell Lung Cancer(NSCLC)
Acronym: BLOSSOM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Se-Hoon Lee, Coordinating investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-09-013
Record Dates: First submitted 2020-09-14; First posted 2020-09-25 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: 80 mg Osimertinib
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 80mg Osimertinib (Experimental): One tablet of 80mg Osimertinib for oral administration per day
  Interventions: Drug: 80mg Osimertinib

INTERVENTIONS:
Drug: 80mg Osimertinib — One tablet of 80mg Osimertinib for oral administration per day
  Other Names: Tagrisso 80mg

SUMMARY:
This will be a Phase II, open-label, single-arm, multicenter study of the efficacy and safety of osimertinib (80 mg orally once daily) in patients with LM associated with EGFRm+ NSCLC.

DETAILED DESCRIPTION:
The study will be conducted in approximately 5 sites across South Korea and will include EGFR TKI pre-treated patients. All patients will be required to have NSCLC associated with at least 1 site of LM as identified by the Investigator that can be assessed by magnetic resonance imaging (MRI) scan and that is suitable for repeat assessments. Presence of Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) measurable intracranial (INC) metastases (ie, brain parenchyma and cranial leptomeninges) and/or extracranial (EXC) metastases is not mandatory. The presence of LM will be based on the Investigator assessment of the brain MRI scan. LM will be confirmed by radiologist from the central site to ensure that patients enrolled in the study are assessable for LM radiologically. Patients negative for LM according to radiologist assessment but enrolled in the study will be replaced. The replaced patient will be included in the study and will receive investigational product (IP) if, in the opinion of the Investigator, the patient is able to receive clinical benefit. Such a patient will not be evaluable for LM response in the LM-EFR analysis set.Full analyses set (FAS) is defined as patients enrolled who received at least 1 dose of study treatment. In addition to Response Assessment in Neuro-Oncology criteria for Leptomeningeal Metastases (RANO-LM) assessments, separate RECIST 1.1 imaging assessments on EXC disease and INC (both LM and non-LM) disease will be performed on images acquired using the preferred method of contrast-enhanced computed tomography (CT) scan of the chest and abdomen (and pelvis when indicated) (EXC) and gadolinium contrast-enhanced MRI scan of the brain (INC).

Baseline scans will be acquired within 28 days prior to first dose of IP and then every 8 weeks (±1 week) and every 12 weeks (±1 week) after 12 months relative to first dose. Patients who discontinue IP for reasons other than objective disease progression in all of INC, EXC, and LM, will continue scans every 8 weeks (±1 week; relative to date of first dose of IP) and every 12 weeks (±1 week, after 12 months) until objective progression in INC, EXC, and LM or withdrawal of consent. Progression refers to progression assessed objectively by imaging using RECIST 1.1 for non-LM INC and EXC or RANO-LM criteria as appropriate. If a patient has been deemed to have LM subjective disease progression according to radiological and clinical assessment by the Investigatorstudy treatment can be continue, and the patient should maintain tumor imaging assessments according to the schedule of assessments.

CSF sampling for cytology is not mandatory, but is strongly encouraged, in patients who are willing to have lumbar punctures during the study, or in those patients who have Ommaya reservoirs.

Physical examination, Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance status score, vital signs, and laboratory tests (hematology, clinical chemistry, and urinalysis) will be conducted at each visit. Adverse events (AEs) will be monitored and recorded on an ongoing basis. Twelve-lead electrocardiograms (ECGs) will be performed at baseline and at the time point of investigator's decision and will include measurement of the QT interval. A multigated acquisition scan (MUGA) or echocardiogram will be performed at baseline and at the time point of investigator's decision for left ventricular ejection fraction (LVEF) measurement. Plasma and CSF (if feasible) samples for pharmacokinetic (PK) analysis will be collected at pre-dose on Cycle 3 Day 1 and Cycle 6 Day 1.

Patient-Reported Outcome (PRO) questionnaires, including European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 items (EORTC QLQ-C30), EORTC Quality of Life Questionnaire-Brain Cancer Module 20 items (EORTC QLQ-BN20) will be collected at baseline (prior to first dose of IP and prior to all other assessments on Cycle 1 Day 1) and at home (every 8 weeks [±3 days for EORTC QLQ-C30 and EORTC QLQ-BN20 relative to administration of IP). The patient is asked to report PROs up to the end of Cycle 8 or to IP discontinuation, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Provision of signed and dated written ICF prior to any mandatory study specific procedures, sampling, and analyses.
3. Male and female patients must be at least 18 years of age.
4. Patients must have documented (only allowed for EGFRm+ [exon 19 deletions or L858R] in pre-treated patients) and/or confirmed central/local test result showing eligible EGFR mutation status as specified below:

   - EGFR TKI pre-treated patients: EGFRm+ (exon 19 deletions or L858R), along with valid T790M mutation status
5. All patients will be required to have NSCLC associated with at least 1 site of LM as identified by the Investigator that can be assessed by MRI scan and that is suitable for repeat assessments. Measurable INC or EXC disease by RECIST 1.1 is not required. Concomitant brain metastases and brain metastases previously treated with radiation therapy are allowed. In addition, asymptomatic untreated BM is also allowed.
6. EGFR TKI pre-treated patients must have had at least 1 prior EGFR TKI (eg, gefitinib, erlotinib, icotinib, dacomitinib or afatinib) and may have had other lines of therapy
7. If the patients is T790M negative, EXC must be stable following previous EGFR TKI treatment. EXC progression is allowed if patients are T790M positive patients
8. ECOG/WHO performance status 0 to 2 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
9. Females must be using highly effective contraceptive measures and must have a negative pregnancy test prior to start of dosing if of childbearing potential, or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:

   * Post-menopausal, defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
   * Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution
   * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation Further information is in Appendix I (Definition of women of childbearing potential and acceptable contraceptive methods).
10. Male patients must be willing to use barrier contraception
11. For inclusion in the optional genetics research study, patients must provide informed consent for genetic research.
12. If a patient declines to participate in any voluntary exploratory research of the study, there will be no penalty or loss of benefit to the patient and he/she will not be excluded from other aspects of the study.

Exclusion Criteria:

1. EGFR TKI pre-treated patients whose T790M mutation status cannot be determined.
2. EGFR TKI pre-treated patients with progressing EXC disease who are T790M mutation-negative. Progressing EXC disease is defined as RECIST 1.1 PD no more than 3 months prior to enrollment, per Investigator assessment.
3. Past medical history of ILD, drug-induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD.
4. Significant medical or psychiatric illness that would interfere with compliance and ability to tolerate treatment as outlined in the protocol.
5. Any of the following cardiac criteria:

   * Mean resting corrected QTc >470 msec, obtained from ECGs, using the screening clinic ECG machine-derived QTc value
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG (eg, complete left bundle branch block, third degree heart block, and second degree heart block)
   * Patients with any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as the following electrolyte abnormalities, heart failure, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes (TdP):

     * Hypokalemia (serum potassium <3.5 mmol/L)
     * Hypomagnesemia (serum magnesium <0.7 mmol/L)
     * Hypocalcemia (corrected serum calcium <2.1 mmol/L)
6. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   * Absolute neutrophil count <1.5×109/L
   * Platelet count <100×109/L
   * Hemoglobin <90 g/L
   * Alanine aminotransferase (ALT) >2.5× the upper limit of normal (ULN) if no demonstrable liver metastases or >5× ULN in the presence of liver metastases
   * Aspartate aminotransferase (AST) >2.5× ULN if no demonstrable liver metastases or >5× ULN in the presence of liver metastases
   * Total bilirubin (TBL) >1.5× ULN if no liver metastases or >3× ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases
   * Creatinine >1.5× ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5× ULN
7. Known INC hemorrhage that is unrelated to tumor.
8. Patients with the clinical manifestation of nervous system failure including severe encephalopathy or with severe nervous system injury related with treatment, such as chemical meningitis.
9. Non-malignant neurological disease that would interfere with evaluation of symptoms or signs of LM.
10. CNS complications that require urgent neurosurgical intervention (eg, resection or shunt placement) up to 2 weeks before to start of IP or patients who have not recovered from side effects of such intervention.
11. Treatment with any of the following:

    * Any cytotoxic chemotherapy, investigational agents, or anticancer drugs (other than EGFR TKI) for the treatment of advanced NSCLC from a previous treatment regimen or clinical study up to 14 days before the first dose of IP.
    * Treatment with an EGFR TKI (eg, afatinib, erlotinib, icotinib, dacomitinib or gefitinib) up to 8 days or approximately 5× half-life, whichever is the longer, before the first dose of IP (if sufficient wash-out time has not occurred due to schedule or PK properties, an alternative appropriate wash-out time based on known duration and time to reversibility of drug-related AEs could be agreed upon by principal investigator).
    * Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of cytochrome P450 (CYP) 3A4 (at least 3 weeks prior) (see Appendix H). All patients must try to avoid concomitant use of any medications, herbal supplements, and/or ingestion of foods with known inducer effects on CYP3A4.
    * Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2 prior platinum-therapy related neuropathy.
    * Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardize compliance with the protocol, or active infection including hepatitis B, hepatitis C, and human immunodeficiency virus. Screening for chronic conditions is not required.
    * Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of osimertinib.
    * Major surgery (excluding placement of vascular access) up to 4 weeks before the first dose of IP.
    * Radiotherapy, as specified, during the following windows:

      * Radiotherapy with a wide field of radiation (including whole brain radiotherapy) up to 2 weeks before the first dose of IP
      * Radiotherapy with a limited field of radiation for palliation up to 1 week before the first dose of IP except for patients receiving radiation to more than 30% of the bone marrow, which must be completed up to 2 weeks before the first dose of IP.
    * Patients receiving intrathecal chemotherapy up to 2 weeks before the first dose of IP.
    * Previously treated with osimertinib.
    * Any requirement for concurrent therapy including radiotherapy for LM other than the specified treatment in this study.
    * Use of corticosteroid to control increased intracranial pressure is allowed
12. History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib.
13. Patient with involvement in the planning and/or conduct of the study (applies to both principal investigator and/or staff at the study site).
14. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
15. Patient has previously participated in the present study, except for rescreened patients with T790M mutation-negative disease who were previously screened but were excluded due to progressing EXC disease that has subsequently been stabilized.
16. For female patients only - Women who are breastfeeding or currently pregnant (confirmed with positive pregnancy test).
17. Contraindication to MRI, including, but not limited to, claustrophobia, pacemakers, metal implants, INC surgical clips, and metal foreign bodies.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 30 months
  To investigate the efficacy of osimertinib on LM as measured by OS

SECONDARY OUTCOMES:
LM ORR(Objective response rate) | Up to 30 months
  BICR(Blinded independent central review) assessments, based on neuroimaging RANO-LM
LM DoR(Duration of response) | Up to 30 months
  BICR(Blinded independent central review) assessments, based on neuroimaging RANO-LM
LM DCR(Disease control rate) | Up to 30 months
  BICR(Blinded independent central review) assessments, based on neuroimaging RANO-LM
LM PFS(Progression-free survival) | Up to 30 months
  BICR(Blinded independent central review) assessments, based on neuroimaging RANO-LM
CSF response rate based on CSF cytology | Up to 30 months
  To investigate the efficacy of osimertinib in patients with LM associated with EGFRm+ NSCLC on the CSF cytological clearance

CONTACTS AND LOCATIONS:
Overall Officials: Se-Hoon Lee, M.D, Ph.D., Principal Investigator — Samsung Medical Center
Locations (6):
- South Korea (6):
  - ChungBuk National University Hospital, Cheonju
  - National Cancer Center, Goyang
  - Seoul National University Bundang Hospital, Seongnam
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park S, Baldry R, Jung HA, Sun JM, Lee SH, Ahn JS, Kim YJ, Lee Y, Kim DW, Kim SW, Lee KH, Lee WJ, Choi JW, Chong K, Lee JI, Gwon SH, Son NH, Ahn MJ. Phase II Efficacy and Safety of 80 mg Osimertinib in Patients With Leptomeningeal Metastases Associated With Epidermal Growth Factor Receptor Mutation-Positive Non-Small Cell Lung Cancer (BLOSSOM). J Clin Oncol. 2024 Aug 10;42(23):2747-2756. doi: 10.1200/JCO.24.00708. Epub 2024 Jun 3. PMID 38828959